CLINICAL TRIAL: NCT01754610
Title: Strengthening Family Coping Resources Open Trials
Acronym: SFCR
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Laurel J Kiser, Prinicipal Investigator; Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00040466
Record Dates: First submitted 2012-12-14; First posted 2012-12-21 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Intervention Effectiveness; Practice-based Evidence; Posttraumatic Stress Disorder
Keywords: family trauma; multi-family therapy; Posttraumatic Stress Disorder; poverty
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Families participating in SFCR: Families who have experienced multiple traumas and high stress related to poverty
  Interventions: Behavioral: Strengthening Family Coping Resources (SFCR)

INTERVENTIONS:
Behavioral: Strengthening Family Coping Resources (SFCR) — Trauma Version (15 weeks) and High Risk Version (10 weeks) are 2 hour sessions. Dinner will be provided at the start of group for all participants.
  Activities will be conducted at each group to encourage family involvement. The treatment modules focus on family rituals and routine, strengthening families' collaborative coping, and resolution of the trauma(s) bringing the families to treatment. Activities will be both family-based and age-based.

SUMMARY:
Strengthening Families Coping Resources (SFCR) Open Trials completes the second stage of the National Institute on Drug Abuse's intervention development model by testing a new family, skills-based intervention involving pre-post evaluation of families participating in multi-family groups. The purpose of this study is to gather practice-based evidence on the effectiveness of the manualized treatment, on the dynamics involved in the group format, and on implementation fidelity and feasibility. Analyses will involve initial exploration of the following hypotheses: 1) Families will show a significant increase in the constructive use of family coping skills and in general family functioning. 2) The target child will show a reduction in trauma-related symptoms and behavior problems. 3) Parents will show significant reductions in traumatic stress and other symptoms of distress. 4) Families will engage and participate in the treatment. 5) Providers will implement SFCR with fidelity.

Other outcomes of interest are the process measures that will be collected to monitor participation in the groups, cultural sensitivity and acceptability, clinician competence, and intervention integrity.

DETAILED DESCRIPTION:
Strengthening Family Coping Resources (SFCR) is a manualized, trauma-focused, skills-based intervention that uses a multi-family group format. SFCR is designed for families living in traumatic contexts with the goal of reducing the symptoms of posttraumatic stress disorder (PTSD) and other trauma-related disorders in children and adult caregivers. Since most families living in traumatic contexts contend with on-going stressors and threats, SFCR is also designed to increase coping resources in children, adult caregivers, and in the family system to prevent relapse and re-exposure. SFCR provides trauma treatment within a family format. SFCR includes additional therapeutic strategies designed to improve the family's ability to cope with on-going stress and threats of re-exposure. Specifically, SFCR builds the coping resources necessary to help families boost their sense of safety, function with stability, regulate their emotions and behaviors, and improve communication about and understanding of the traumas they have experienced. The model includes family work on storytelling and narration, which builds to a family trauma narrative. SFCR is currently being implemented at University of Maryland Medical Center (UMMC), at sites that are part of the National Child Traumatic Stress Network (NCTSN), and at community agencies within the Baltimore Metro area and beyond.

Families will participate in a multifamily version of the intervention. Multiple groups of 5-6 families will be conducted with pre-post data collected in addition to information on the feasibility of the intervention. Prior to beginning each group, families will be assessed using a structured assessment. This assessment will be repeated at the end of group (all groups) and approximately one year following the completion of the group (for UMMC groups only).

One child in each family will be designated as the research subject. The target child will be chosen according to age, aged 1 through 17 years old, and referral for services. If more than one child in the family meet these criteria, the primary caregiver will be given the option of how many children s/he would like to be assessed for inclusion in the study. Data on the parents will only be collected from mothers or female caregivers. If no female caregiver is available, the primary caregiver will complete the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 through 17 years old at the time of recruitment
* Child and family exposed to multiple traumas
* a partial diagnosis of PTSD (15-week treatment version)
* currently in the custody of a caregiver who agrees to participate in the study.
* a stable caregiving system as defined by a recent history of stability and unlikely to change in the next 6 months.

Exclusion Criteria:

* Children will be excluded only if they have active suicide ideation, an imminent risk for re-exposure due to their living environment, active psychosis, severe mental retardation or brain injury
* Parent/caregiver has active psychosis or is a danger to self/others.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-02; Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Pre-post Treatment Effects | Change from baseline to end of 10 or 15 week group and 3 month follow up
  This is a large open-ended sample involving collection of practice-based evidence of intervention effectiveness related to broad dissemination. The sample size is not being constrained by a specific research question.
  Data analysis: Indications of change were assessed using pre-post measures. Post-intervention change will be assessed with t-tests for dependent samples. Cohen's d will be used to calculate effect size. Comparison of pre-post scores for the target child will be assessed on PTSD symptoms (UCLA-PTSD Reaction Index Parent and Child Versions) and on behavior problems (CBCL). Comparison of pre-post scores on standardized measures of family functioning (Family Assessment Device), family coping (F-COPES), and parental stress (PSI_SF), and scores on the Family Mealtime Q-Sort will be made.
McMaster Family Assessment Device (FAD) or General Functioning Scale (FAD 12) | Change from baseline to end of 10 or 15 week group and 3 month follow up
  The McMaster Family Assessment Device (FAD) (Epstein et al., 1983; Miller, Epstein, Bishop, & Keitner, 1985) is a 60-question, Likert scale instrument designed to measure family functioning based upon the McMaster Model. Items are scored on a 4-point scale from 1 "healthy" to 4 "unhealthy." The instrument provides scores for seven scales, including problem-solving, communication, roles, affective responsiveness, affective involvement, behavior control, and overall functioning.
Child Behavior Checklist (CBCL) | Change from baseline to end of 10 or 15 week group and 3 month follow up
  Providers of SFCR can choose to administer 1 of 3 measures of behavior problems in children. The CBCL/1½-5 and 6-18 (Achenbach & Rescorla, 2001) requires a caregiver to rate, on a three-point scale from 0 (not true) to 2 (often true), each of 118 problems as they are perceived to reflect the child's behavior over the past six months. The instrument has 8-9 subscales that can be collapsed into broadband scales: Internalizing, Externalizing, and a Total Score.
UCLA PTSD Reaction Index | Change from baseline to end of 10 or 15 week group and 3 month follow up
  This instrument measures exposure to and symptoms of trauma in school-age children and adolescents. Symptoms assessed are tied to Diagnostic and Statistical Manual criteria for Posttraumatic Stress Disorder (PTSD). The UCLA PTSD-RI can be used as either a self-report or clinician-administered instrument. Reliability and validity are fairly robust (Steinberg et al., 2004). It has been used in many research designs and, importantly for the purposes of this study, among children exposed to community stress and violence.
Pediatric Symptom Checklist (PSC 17) | Change from baseline to end of 10 or 15 week group and 3 month follow up
  Providers of SFCR can choose to administer 1 of 3 measures of behavior problems in children. The PSC is a short 17-item measure of internalizing and externalizing behaviors.
Strengths and Difficulties Questionnaire (SDQ) | Change from baseline to end of 10 or 15 week group and 3 month follow up
  Providers of SFCR can choose to administer 1 of 3 measures of behavior problems in children. The SDQ is a short measure of child strengths and difficulties and includes indices of internalizing and externalizing problems.
Family Crisis Oriented Personal Evaluation Scales (F-Copes) | Change from baseline to end of 10 or 15 week group and 3 month follow up
  Inventory that measures family coping.

SECONDARY OUTCOMES:
Parent Symptoms of PTSD | Change from baseline to end of 10 or 15 week group
  Measured using the PTSD Checklist for DSM-5, a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD (Blevins, Weathers, Davis, Witte, & Domino, 2015). The PCL-5 was developed to assess symptom change during and after treatment, to screen for clinically significant PTSD symptoms, and to make provisional PTSD diagnoses.
Parent General Symptoms | Change from baseline to end of 10 or 15 week group
  Brief Symptom Inventory-18 item (BSI) (Derogatis, 2000) is an 18-item self-report inventory of adult (18 years and older) psychological symptoms.

OTHER OUTCOMES:
SFCR Facilitator Competence and Fidelity | Completed after each session
  These are short self-report measures of each facilitators' impressions of their competence during the group and their adherence to the session guidelines.
Family Feedback and Satisfaction Forms | Completed after each session and at the beginning and ending of SFCR
  Forms that provide family impressions of SFCR.

CONTACTS AND LOCATIONS:
Overall Officials: Laurel J Kiser, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, School of Medicine, Department of Psychiatry, Divsion of Services Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiser LJ, Donohue A, Hodgkinson S, Medoff D, Black MM. Strengthening family coping resources: the feasibility of a multifamily group intervention for families exposed to trauma. J Trauma Stress. 2010 Dec;23(6):802-6. doi: 10.1002/jts.20587. PMID 21105068
- [Background] Kiser LJ, Baumgardner B, Dorado J. Who Are We, But for the Stories We Tell: Family Stories and Healing. Psychol Trauma. 2010 Sep 1;2(3):243-249. doi: 10.1037/a0019893. PMID 21197420
- [Background] Kiser, LJ., Backer, PM., Winkles, JK., Medoff, D. Strengthening Family Coping Resources (SFCR): Practice-Based Evidence for a Promising Trauma Intervention. Couple and Family Psychology: Research and Practice 4:49-59, 2015. Doi:10/1037/cfp0000034
- [Background] Kiser, LJ, Miller, AB, Mooney, MA, Vivrette, R, Davis, S. Integrating parents into child trauma treatment: Reviewing evidence and establishing core components. Practice Innovations. 2020; 5:65-80. doi: http://dx.doi.org/10.1037/pri0000109